CLINICAL TRIAL: NCT07341945
Title: Association Between Oral Health Literacy and Periodontal Status Among Turkish Adults: A Cross-Sectional Study
Brief Title: Oral Health Literacy and Periodontal Status Among Turkish Adults
Status: Completed | Type: Observational
Sponsor: Biruni University (Other)
Responsible Party: Principal Investigator, Burcu KARADUMAN, Principal Investigator, Biruni University
Other Study IDs: 2024-BİAEK/12-14; 2024-BIAEK/12-14 (Other: Biruni University Non-Interventional Ethics Committee (Istanbul, Türkiye))
Record Dates: First submitted 2026-01-06; First posted 2026-01-15 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2026-01

CONDITIONS: Periodontal Diseases; Oral Health Literacy; Periodontitis; Health Behaviour; Health Education
Keywords: Periodontitis, Health Behaviour, Oral Hygiene, Socioeconomic Status, Health Education, Smoking.
MeSH Terms: conditions — Periodontal Diseases; Periodontitis; Health Education; Smoking

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Adult Participants: A single observational group including adult individuals who attended Biruni University Faculty of Dentistry, Istanbul, Türkiye. All participants underwent a full-mouth periodontal examination and completed the Turkish version of the Rapid Estimate of Adult Literacy in Dentistry (TREALD-30) questionnaire. No intervention or treatment was provided as part of the study.
  Interventions: Other: Observational Assessment

INTERVENTIONS:
Other: Observational Assessment — No intervention was performed. Participants underwent a non-invasive periodontal examination and completed the Turkish version of the Rapid Estimate of Adult Literacy in Dentistry (TREALD-30) questionnaire to assess oral health literacy.

SUMMARY:
This observational cross-sectional study aimed to investigate the association between oral health literacy (OHL) and periodontal status among adult individuals attending Biruni University Faculty of Dentistry, Istanbul, Türkiye. A total of 108 adults were evaluated using the Turkish version of the Rapid Estimate of Adult Literacy in Dentistry (TREALD-30) to assess OHL levels. Periodontal examination included probing depth, clinical attachment level, bleeding on probing, and plaque index. The study sought to determine whether lower OHL levels are associated with poorer periodontal health and to highlight the importance of improving health literacy in oral disease prevention and management.

DETAILED DESCRIPTION:
This cross-sectional observational study was conducted at Biruni University Faculty of Dentistry, Istanbul, Türkiye, to evaluate the relationship between oral health literacy (OHL) and periodontal status among adult individuals. A total of 108 systemically healthy adults aged 18 years or older were included. Individuals with fewer than 20 teeth, history of periodontal treatment in the past 6 months, or systemic diseases affecting periodontal health were excluded.

OHL was assessed using the validated Turkish version of the Rapid Estimate of Adult Literacy in Dentistry (TREALD-30). Periodontal examination was performed by a calibrated periodontist and included full-mouth probing depth (PD), clinical attachment level (CAL), bleeding on probing (BOP), and plaque index (PI). Periodontitis was defined according to the 2018 World Workshop classification system.

The primary objective was to determine whether limited OHL is associated with worse periodontal parameters. Secondary objectives included evaluating the relationship between OHL and sociodemographic variables such as age, education, and smoking habits. Statistical analyses were performed using regression models to identify independent predictors of periodontal disease.

The findings of this study aim to emphasize the role of oral health literacy as a potential social determinant of periodontal health and to guide the development of literacy-based preventive strategies in dental public health.

ELIGIBILITY:
Inclusion Criteria:

Systemically healthy adults aged 18 years or older

Ability to read and understand Turkish

Voluntary agreement to participate in the study

Exclusion Criteria:

Individuals with fewer than 20 teeth

History of periodontal treatment within the past 6 months

Presence of systemic diseases affecting periodontal health

Individuals with mental retardation, cognitive impairment, or inability to complete the questionnaire due to illiteracy or communication difficulties

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study included 108 systemically healthy adults aged 18 years or older who attended the Periodontology Clinic of Biruni University Faculty of Dentistry, Istanbul, Türkiye. Participants were native Turkish speakers, able to read and understand Turkish, and provided informed consent. Each participant completed the Turkish version of the Rapid Estimate of Adult Literacy in Dentistry (TREALD-30) to assess oral health literacy. Periodontal examinations were performed by a calibrated periodontist and included probing depth, clinical attachment level, bleeding on probing, and plaque index measurements. Individuals with systemic diseases, fewer than 20 teeth, or cognitive or literacy limitations preventing questionnaire completion were excluded.
Sampling Method: Non-Probability Sample
Enrollment: 108 (Actual)
Dates: Start 2021-09-01 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2024-07-31 (Actual)

PRIMARY OUTCOMES:
Association between oral health literacy and periodontal status | Baseline (single examination at enrollment)
  The primary outcome is the relationship between oral health literacy, measured by the Turkish version of the Rapid Estimate of Adult Literacy in Dentistry (TREALD-30), and periodontal status based on the 2018 World Workshop classification. Periodontal parameters include probing depth (PD), clinical attachment level (CAL), and bleeding on probing (BOP).

SECONDARY OUTCOMES:
Association between oral health literacy and demographic factors | Single time point (baseline examination)
  To assess the association between oral health literacy levels and demographic characteristics such as age, gender, and educational attainment among adult participants.
Relationship between oral health literacy and smoking status | Single time point (baseline examination)
  To determine whether smoking habits are associated with lower oral health literacy scores and poorer periodontal parameters.
Association between oral health literacy and oral hygiene behaviors | Single time point (baseline examination)
  To evaluate the relationship between oral health literacy (measured by the TREALD-30) and self-reported oral hygiene practices, including toothbrushing frequency, use of interdental cleaning aids, and frequency of dental visits.

CONTACTS AND LOCATIONS:
Overall Officials: Burcu Karaduman, DDS, PhD, Study Director — Biruni University Faculty of Dentistry
Locations (1):
- Biruni University Faculty of Dentistry, Department of Periodontology, Istanbul, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be shared because this observational study involves identifiable clinical and questionnaire data collected under institutional ethics approval, which restricts public data sharing due to privacy and confidentiality considerations.